CLINICAL TRIAL: NCT06636422
Title: Post-marketing Safety and Efficacy Surveillance of Motherwort Injection : a Registry Study
Brief Title: Post-marketing Safety and Efficacy Surveillance of Motherwort Injection
Status: Not yet recruiting | Type: Observational
Sponsor: Zhong Wang (Other)
Responsible Party: Sponsor-Investigator, Zhong Wang, Sponsor, China Academy of Chinese Medical Sciences
Organization: China Academy of Chinese Medical Sciences (Other)
Other Study IDs: Motherwort-V2.0
Record Dates: First submitted 2024-09-30; First posted 2024-10-10 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-03

CONDITIONS: Bleeding; Real-world Study; Adverse Events
Keywords: Adverse events; Motherwort injection; bleeding; real-world study; Post-abortion hemorrhage; Uterine retraction
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients indicated for Motherwort injection: During the registration and enrollment period of the study, all patients who meet the clinical indications for the use of motherwort injection, as determined by the physician, and voluntarily agree to participate while fulfilling ethical requirements, will be recruited from designated medical institutions and departments. The observation period for each observer was established based on the clinical application of motherwort injection.
  Interventions: Drug: Motherwort injection

INTERVENTIONS:
Drug: Motherwort injection — Patients will be given motherwort injection according to their disease condition in the real world. The investigator only can record the information on the usage of the drug and the relevant medications without any interventions.
  Other Names: Yimucao Injection

SUMMARY:
This study aims to provide evidence concerning the safety and efficacy of motherwort injection in real-world settings.

ELIGIBILITY:
Inclusion Criteria:

* Meet the clinical indications for the use of motherwort injection
* Voluntarily participate in this study
* Fulfill ethical requirements.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients from designated medical institutions (departments) who meet the clinical indications for the use of motherwort injection as determined by a physician, voluntarily participate in this study, and fulfill ethical requirements.
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2024-10-15 (Estimated); Primary Completion 2025-10-15 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
The type and incidence of adverse events. | From the initiation of medication to 7 days after cessation.
Bleeding control. | From the commencement of the surgery to the end of bleeding event, assessed up to 1 year.
  Including:1. Hysteroscopic surgery: the intraoperative blood loss, the postoperative blood loss, the cumulative bleeding time.
  2.Uterine fibroid resection: the intraoperative blood loss, the postoperative blood loss, the cumulative bleeding time.
The incidence of postpartum hemorrhage. | From the completion of the surgery to 24 hours following the delivery of the fetus.
  Postpartum hemorrhage is defined as a blood loss of ≥500 ml following vaginal delivery or ≥1000 ml following cesarean delivery, or the presence of symptoms or signs of hypovolemia associated with blood loss within 24 hours .
The post-abortion recovery. | From the completion of the abortion to the subsequent onset of menstruation, assessed up to 1 year.
  The interval time to the resumption of menstruation post-surgery.
The incidence of post-abortion bleeding. | From the completion of the abortion to the end of bleeding event.
  The cumulative days of postoperative bleeding.

SECONDARY OUTCOMES:
The types and incidence of adverse reactions. | From the initiation of medication to 7 days after cessation.
Analysis of factors associated with adverse reactions. | From the initiation of medication to 7 days after cessation.
The menstrual adjustment. | From the initiation of medication to menstruation returns to normal or the treatment is completed, whichever came first, assessed up to 1 year.
  Ovulatory dysfunction-related abnormal uterine bleeding: utilizing a treatment satisfaction assessment (0 = dissatisfied; 1 = neutral; 2 = somewhat satisfied; 3 = very satisfied).
The uterine retraction status. | From the the postpartum to the end of bleeding event, assessed up to 1 year.
  Including:1.Rate of poor uterine involution: poor uterine involution is defined as the persistence of lochia beyond 42 days postpartum. 2. Duration of lochia cessation.

OTHER OUTCOMES:
The assessment of treatment satisfaction. | From the initiation of medication to 7 days after cessation.
  A four-level rating scale was employed, as follows: 0 = dissatisfied; 1 = neutral; 2 = somewhat satisfied; 3 = very satisfied.